CLINICAL TRIAL: NCT03259854
Title: Non Invasive Mechanical Ventilation VERSUS Oxygen MASK After Successful Weaning From Invasive Mechanical Ventilation in Pediatrics
Brief Title: Non Invasive Mechanical Ventilation VERSUS Oxygen MASK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Khalaf, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NVM
Record Dates: First submitted 2017-08-13; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Mechanical Ventilation Complication
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxygen mask control group (Active Comparator): patients will receive oxygen by mask will be monitored regarding oxygen saturation, blood pressure, respiratory rate, heart rate, arterial blood gases
  Interventions: Device: oxygen mask
- non invasive ventilation study group (Experimental): patients will receive non invasive ventilation after successful weaning from invasive ventilation and will be monitored regarding oxygen saturation, blood pressure, respiratory rate, heart rate, arterial blood gases
  Interventions: Device: non invasive mechanical ventilation in pediatrics

INTERVENTIONS:
Device: non invasive mechanical ventilation in pediatrics — use of non invasive mechanical ventilation in pediatrics after successful weaning from invasive mechanical ventilation
  Arms: non invasive ventilation study group
Device: oxygen mask — use of oxygen mask after successful weaning from invasive mechanical ventilation
  Arms: oxygen mask control group

SUMMARY:
Conventional mechanical ventilation is a core feature of intensive care. Weaning and removal of endotracheal tube are crucial processes, which often account for a considerable part of Conventional mechanical ventilation total time. Unsuccessful extubation has been noted to be associated with an increase of both morbidity and mortality in adult and pediatric patients

DETAILED DESCRIPTION:
The documented rate of failed extubations ranges from 4.1 to 14% in pediatric intensive care units.Therefore, strategies preventing the need for reintubation are needed.

Non invasive ventilation has been proposed as useful therapy to wean patients after unsuccessful weaning trials and to avoid reintubation in adults, though controversy exists at this concern.

This technique is increasingly being used in pediatric patients over the last years. The objective of the present study was to determine post extubation Non invasive ventilation characteristics and to identify risk factors of post extubation Non invasive ventilation failure in children

ELIGIBILITY:
Inclusion Criteria:

all the patients with successful weaning from invasive mechanical ventilation

Exclusion Criteria:

1. Maxillofacial trauma
2. Gastrointestinal obstruction
3. Severe lung secretion
4. Irreversible organ failure

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
risk of respiratory failure after non invasive ventilation use | one week after successful weaning from invasive mechanical ventilation
  The patients will be evaluated to determine any manifestation of respiratory failure

SECONDARY OUTCOMES:
complications of non invasive mechanical ventilation in pediatrics | one week after use of non invasive ventilation
  monitor any complications from use of Non Invasive Ventilation
length of hospital stay after non invasive ventilation use | one month after use of non invasive ventilation
  the duration of hospital stay for all patients will be recorded

REFERENCES:
- [Result] Ferrer M, Sellares J, Valencia M, Carrillo A, Gonzalez G, Badia JR, Nicolas JM, Torres A. Non-invasive ventilation after extubation in hypercapnic patients with chronic respiratory disorders: randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1082-8. doi: 10.1016/S0140-6736(09)61038-2. Epub 2009 Aug 12. PMID 19682735
- [Result] Baisch SD, Wheeler WB, Kurachek SC, Cornfield DN. Extubation failure in pediatric intensive care incidence and outcomes. Pediatr Crit Care Med. 2005 May;6(3):312-8. doi: 10.1097/01.PCC.0000161119.05076.91. PMID 15857531
- [Result] Trevisan CE, Vieira SR; Research Group in Mechanical Ventilation Weaning. Noninvasive mechanical ventilation may be useful in treating patients who fail weaning from invasive mechanical ventilation: a randomized clinical trial. Crit Care. 2008;12(2):R51. doi: 10.1186/cc6870. Epub 2008 Apr 17. PMID 18416851